CLINICAL TRIAL: NCT01285024
Title: A Prospective Study to Evaluate the Effectiveness of a Haemostatic Agent in Primary Unilateral Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Orthovita d/b/a Stryker (Industry); Stryker Instruments (Industry)
Responsible Party: Principal Investigator, Wael Barsoum, MD, Chairman of Surgical Operations, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCF 10-916
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Arthritis
Keywords: total hip arthroplasty; transfusion; hemostat
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No Vitagel used during total hip arthroplasty
- Vitagel (Experimental): Vitagel applied just prior to closure during total hip arthroplasty
  Interventions: Device: Vitagel

INTERVENTIONS:
Device: Vitagel — Two 4.5mL Vitagel Surgical Hemostat Kits, used just prior to closing the capsule.
  Arms: Vitagel

SUMMARY:
This is a prospective, randomized, controlled, single-center study to assess the effectiveness of Vitagel, a surgical hemostat, in primary unilateral total hip arthroplasty (THA). This will be an inter-patient controlled study involving one-hundred-ten subjects. Vitagel will be used in a randomly selected cohort of fifty-five patients undergoing primary unilateral THA procedures; a control group of fifty-five patients will not receive Vitagel or any other hemostatic agent except those that are standard during a primary THA. The study will evaluate the effectiveness of Vitagel in reducing intra- and post-operative bleeding.

DETAILED DESCRIPTION:
Vitagel Surgical Hemostat is composed of microfibrillar collagen and thrombin in combination with autologous plasma. It is applied to the surgical site as a sprayable liquid which then forms a collagen/fibrin gel matrix (containing the patients activated platelets) which adheres to the bleeding site. This matrix provides hemostasis and facilitates healing. Vitagel is resorbed in approximately 30 days. It is easily prepared by the OR staff in minutes and only requires ~10mL's of the patient's blood per Vitagel 4.5ml kit. Compared to other hemostatic agents on the market today, Vitagel has the advantages of not containing pooled human donor blood proteins, aprotinin, or tranexamic acid.

Vitagel has been studied in multiple surgical specialties to demonstrate safety and efficacy. Vitagel was studied in orthopedic procedures, both on iliac crest donor sites and sternal edges, during its IDE studies for FDA approval. Vitagel was granted broad indications for use by the FDA in 2000 as an adjunct to hemostasis. It was formerly marketed under the name CoStasis® Surgical Hemostat, by Cohesion Technologies, Palo Alto, CA.

The use of a surgical hemostat in joint arthroplasty may substantially decrease post-operative blood loss, which may reduce patient morbidity, length of hospital stay, and costs by potentially eliminating the need for transfusions and drains.

Total Hip Arthroplasty (THA) is associated with post-operative blood loss and frequently requires the transfusion of blood products. Increased concern over the risks of blood transfusion, which include transmission of viral diseases, such as HIV, Hepatitis, and CMV as well as transfusion reactions, has perpetuated the search for new methods of blood conservation in orthopedic surgery. There exists considerable variation in the protocols that are used to optimize hemostasis and minimize post-operative blood loss in patients undergoing THA. Some methods used include pre-operative hemodilution and hypotensive anesthesia; however, these methods have associated risks, require careful monitoring, and can prolong the operative time. Another method used is intra-operative and post-operative salvage of blood with re-infusion which requires continuous monitoring and is limited to patients who bled heavily during the initial period following surgery, because the blood should be collected over a period of not more than six hours. The transfusion of autologous pre-donated blood is also commonly used in THA surgery. While autologous pre-donated blood is not associated with the risk of viral disease transmission, the rates of administrative error and bacterial overgrowth (the factors most frequently associated with immediate post-transfusion deaths) are comparable with those associated with the use of homologous blood. The collection of pre-donated blood requires special programs and scheduling. Studies have indicated that the use of autologous blood transfusions may have little health benefit at considerable costs.

During surgery, meticulous electrocautery, helps minimize both acute blood loss and post-operative drainage. No uniform guidelines exist regarding the use of post-operative drains in THA. Some surgeons use drain systems that allow re-infusion of the erythrocytes, others prefer simple vacuum drains. Still others do not use drains at all. There are conflicting data regarding the efficacy of closed suction drains. Some studies have shown that bleeding may be potentiated by suction drainage. Other studies have shown that drains can lead to complications such as infection, increased blood loss, need for blood transfusions, breakage in the drain tube, and pain during drain tube removal. Thus, the need for adequate hemostasis in THA remains apparent.

To date there have been limited published studies on the use of hemostatic agents during THA procedures. However, even in a relatively low number of patients these studies have shown that the use of hemostatic agents is a safe and effective means to reduce blood loss and the need for and rate of blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled for a primary unilateral THA;
* Are able and willing to provide voluntary written informed consent for participation in the study;
* Are between the ages of 18 and 85 at the time of surgery;
* Are willing to comply with all aspects of the treatment and evaluation period

Exclusion Criteria:

* Are known to be sensitive to any materials of bovine origin;
* Are undergoing a bilateral or revision THA;
* Patients predonating autologous blood.
* Patients with a preoperative platelet count of less than 100,000.
* Patients with a previous history of venous thromboembolism or deep vein thrombosis
* Medical condition requiring anticoagulation
* Currently using Coumadin
* History of Heparin induced thrombocytopenia or Lovenox induced thrombocytopenia
* Have a history of rheumatoid arthritis or inflammatory arthritis;
* Peripheral vascular disease.
* Evidence of bleeding or metabolic - based hemolytic disorder (hemophilia or anticoagulation use), or hypercoaguable disorder.
* Patients with history of liver disease. Patients with liver dysfunction from cirrhosis or hepatitis may have impaired production of factors in the clotting cascade which may make these individuals more prone to bleed, especially with the use of anticoagulants. For this reason, these patients will also be excluded from this study if a baseline INR is greater than 1.3 or APTT greater than 32.4
* Have a history of failed treatment for abuse of, or are actively abusing, illegal drugs, solvents, or alcohol;
* Have a systemic infection or infection at site of surgery;
* Are a prisoner; and/or
* Are pregnant or nursing.
* Condition deemed by physician or medical staff to be non-conducive to patient's ability to complete the study, or a potential risk to the patient's health and well-being.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-12; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wael K Barsoum, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Vitagel
Started | 49 | 60
Completed | 49 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Vitagel | Total
Number analyzed (Participants) | 49 | 60 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.4) | 58.2 (11.8) | 58.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 18 | 27 | 45
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (6.7) | 32.6 (7.0) | 31.5 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Transfusion Requirement
Description: Measure Title: Units of transfusion required
Time Frame: intraoperative - 1 week postoperative
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Control | Vitagel
Number analyzed (Participants) | 49 | 60
units | 1.6 (0.5) | 2.2 (1.3)

2. Secondary Outcome: Total Hemoglobin Level Change
Description: Total hemoglobin level change from preop to postoperative discharge.
Time Frame: day of surgery - 1 week postoperative
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Control | Vitagel
Number analyzed (Participants) | 49 | 60
g/dL | 4.8 (1.1) | 4.6 (1.2)

ADVERSE EVENTS:
Arm/Group | Control | Vitagel
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/60
Other Adverse Events (participants affected / at risk) | 5/49 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=49) | Vitagel (N=60)
PE/DVT (Vascular disorders) | 1 (1) | 1 (1)
Wound drainiage (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=49) | Vitagel (N=60)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary Retention/Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema with pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Dizziness (General disorders) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No